CLINICAL TRIAL: NCT00001462
Title: Characterization of the Pathobiology of Early Lung Destruction in Alpha 1-Antitrypsin Deficient Individuals
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950116; 95-H-0116
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-08

CONDITIONS: Emphysema; Lung Diseases, Obstructive; Alpha 1-Antitrypsin Deficiency
Keywords: Alpha 1-Antitrypsin Deficiency; Emphysema; Genetic Diseases; Inflammation; Nitric Oxide; Protease
MeSH Terms: conditions — Emphysema; Lung Diseases, Obstructive; alpha 1-Antitrypsin Deficiency; Genetic Diseases, Inborn; Inflammation

SUMMARY:
Alpha 1-antitrypsin-deficient individuals develop severe destructive lung disease much earlier and their lung function declines faster than the general population of individuals with chronic obstructive lung disease. This study is designed to better understand the pathogenesis of lung destruction in alpha 1-antitrypsin deficient individuals and to characterize the pathobiology of early lung destruction. To accomplish this we intend to use bronchoalveolar lavage to determine and quantify the factors that initiate and sustain lung inflammation in alpha 1-antitrypsin deficient individuals with lung function above a force expiratory volume in one second (FEV1) of greater than 50% of predicted.

DETAILED DESCRIPTION:
Alpha 1-antitrypsin-deficient individuals develop severe destructive lung disease much earlier and their lung function declines faster than the general population of individuals with chronic obstructive lung disease. This study is designed to better understand the pathogenesis of lung destruction in alpha 1-antitrypsin deficient individuals and to characterize the pathobiology of early lung destruction. To accomplish this we intend to use bronchoalveolar lavage to determine and quantify the factors that initiate and sustain lung inflammation in alpha 1-antitrypsin deficient individuals with lung function above a force expiratory volume in one second (FEV1) of greater than 50% of predicted.

ELIGIBILITY:
Any alpha 1 antitrypsin-deficient individuals.

18-65 years old.

FEV1 greater than 1 equal to 50 percent of predicted (forced expiratory volume).

Study participation is required for one year.

A total of four bronchoscopies will be performed over a year period.

Methacholine challenge test will be performed at the beginning and end of the study to assess the degree of reactive airways disease.

Pneumococcal and annual influenza vaccine will be given.

No prolastin within one year prior to start of the study.

No oral systemic corticosteroids within 30 days prior to start of study.

No allergy to topical or local anesthetic (i.e., lidocaine).

No pregnancy.

No HIV positive patients.

No Hepatitis B/C virus positive patients.

No patients with any condition associated with immunodeficiency.

No patients with presence of significant cardiac diseases.

No patients with presence of uncorrected blood-clotting disorders.

No patients with any oxygen at home on a regular basis.

No adverse reactions to methacholine.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 1995-05; Study Completion 2000-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Buist AS. Alpha 1-antitrypsin deficiency in lung and liver disease. Hosp Pract (Off Ed). 1989 May 15;24(5):51-9. doi: 10.1080/21548331.1989.11703712. No abstract available. PMID 2497126
- [Background] Crystal RG. Alpha 1-antitrypsin deficiency, emphysema, and liver disease. Genetic basis and strategies for therapy. J Clin Invest. 1990 May;85(5):1343-52. doi: 10.1172/JCI114578. No abstract available. PMID 2185272
- [Background] Gadek JE, Pacht ER. The protease-antiprotease balance within the human lung: implications for the pathogenesis of emphysema. Lung. 1990;168 Suppl:552-64. doi: 10.1007/BF02718178. PMID 2117164
- [Derived] Paris AE, Vragovic O, Sonalkar S, Finneseth M, Borgatta L. Mifepristone and misoprostol compared to osmotic dilators for cervical preparation prior to surgical abortion at 15-18 weeks' gestation: a randomised controlled non-inferiority trial. BMJ Sex Reprod Health. 2019 Nov 21:bmjsrh-2019-200367. doi: 10.1136/bmjsrh-2019-200367. Online ahead of print. PMID 31754065